CLINICAL TRIAL: NCT00684073
Title: Evaluation of Preference for a Buprenorphine-based Maintenance Therapy, After a Switch From Buprenorphine Alone (Subutex®) to the Buprenorphine/Naloxone Combination (Suboxone®), in Opioid-dependent Patients With Buprenorphine Maintenance Therapy
Brief Title: Preference for Subutex® (Buprenorphine) Versus Suboxone® (Buprenorphine/Naloxone) in Opioid Dependent Patients on Subutex® (Study P05094)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05094; 2006-006686-17
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2010-01-01 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Opiate-related Disorders; Opiate Dependence; Drug Abuse
Keywords: Suboxone; Subutex; Buprenorphine; Naloxone
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subutex®/Suboxone® (Experimental): Subutex® for first two days of study followed by Suboxone® for last 3 days of study
  Interventions: Drug: buprenorphine; Drug: buprenorphine/naloxone

INTERVENTIONS:
Drug: buprenorphine — 2 mg buprenorphine and 8 mg buprenorphine tablets at doses from 2 to 16 mg buprenorphine daily for first two days of study
  Other Names: Subutex®; SCH 028444
Drug: buprenorphine/naloxone — 2/0.5 mg buprenorphine/naloxone and 8/2 mg buprenorphine/naloxone tablets at doses from 2/0.5 mg buprenorphine/naloxone to 16/4 mg buprenorphine/naloxone daily for last 3 days of study
  Other Names: Suboxone®; SCH 000484

SUMMARY:
This study is designed to determine if opioid dependent subjects who are already receiving Subutex® prefer the Suboxone® tablet over the Subutex® tablet after switching from Subutex® to Suboxone®. Subjects who are selected to participate in this study will continue their prescribed dose of Subutex® (buprenorphine 2 to 16 mg daily) for the first two days of the study (Day 1 and Day 2) then switch to and receive an equivalent dose of Suboxone® (buprenorphine 2 to 16 mg daily) for the last 3 days of the study (Day 3, Day 4 and Day 5). The Day 5 Visit will be the subject's last study visit. Upon completing the study, subjects will continue their pre-study prescribed dosage of Subutex®.

ELIGIBILITY:
Inclusion Criteria:

* Subject must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Subject must be at least (>=) 18 years of age, of either sex.
* Subject treated for opioid dependence with Subutex® with a stable daily dose between 2 mg and 16 mg daily, for at least 6 months.
* Subject who do not inject/misuse their treatment with Subutex®.
* Subject must be free of illicit opiate drug use as assessed by urine test performed prior to inclusion.
* Subject must understand and be able to adhere to the dosing and visit schedules, and agree to report concomitant medications / products and adverse events to the investigator or designee.
* Women of childbearing potential (includes women who are less than one year postmenopausal and women who become sexually active) must be using or agree to use an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterile (e.g., hysterectomy or tubal ligation).
* Women of childbearing potential should be counseled in the appropriate use of birth control while in this study. Women who are not currently sexually active must agree and consent to use one of the above-mentioned methods should they become sexually active while participating in the study. Women of childbearing potential must have a urine pregnancy test with negative result within 2 weeks prior to inclusion (as performed under control of the investigator or designee).

Exclusion Criteria:

* Subject not eligible for treatment with Subutex® or Suboxone® according to the legal drug attachments.
* Subject refusing to take the daily dose of the study medication under control in the center.
* Subject unable to complete the evaluations.
* Women who are pregnant or nursing.
* Subject with a history of hypersensitivity to buprenorphine hydrochloride or naloxone hydrochloride dihydrate or any excipient of Subutex® or Suboxone®.
* Subject with a current evidence of alcohol abuse.
* Subject with severe respiratory dysfunction, severe hepatic dysfunction, acute alcohol intoxication or delirium tremens .
* Subject with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucosegalactose malabsorption.
* Initiation or increase in the dose, within the past 7 days or scheduled during the study, of a treatment with:

  * benzodiazepines,
  * other depressants of the central nervous system: other morphine derivatives (analgesics, antitussives), certain antidepressive agents, sedative H1 antihistamines, barbiturates, benzodiazepines, anxiolytics other than benzodiazepines, neuroleptics, clonidine and clonidine-like agents and monoamine oxidase [MAO] inhibitors,
  * CYP3A4 inhibitors,
  * CYP3A4 inducers.
* Subjects who have any current evidence of clinically significant hematopoietic, metabolic, cardiovascular, immunologic, neurologic, hematological, gastrointestinal, hepatic, renal, psychiatric, cerebrovascular, or respiratory disease, or any other disorder which, in the judgment of the investigator, may interfere with the study evaluations or affect subject safety.
* Subjects who have used any investigational product within 30 days prior to enrollment.
* Subjects participating in another trial at the same time.
* Subject who intend to donate blood during the study or within 3 months after study completion.
* Subjects in the exclusion period of the "Fichier National des Personnes qui se Prêtent à des Recherches Biomédicales" (National Index of Persons Participating in Biomedical Researches, or National Index of Volunteers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 subjects who started selection were the number of subjects who attended the selection visit and signed informed consent
Period: Selection
Arm/Group | Subutex®/Suboxone®
Started | 60
Completed | 53 (number of subjects who had a Day 1 visit)
Not Completed | 7
Not completed — Selection/non-selection criteria | 3
Not completed — Death | 1
Not completed — noncompliance | 1
Not completed — Lost to Follow-up | 1
Not completed — request of the sponsor | 1
Period: Treatment (Days 1 Through 5)
Arm/Group | Subutex®/Suboxone®
Started | 53 (number of subjects who had a Day 1 visit)
Completed | 52 (number of subjects who had a Day 5 visit (and therefore completed study))
Not Completed | 1
Not completed — non-respect of eligibility criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subutex®/Suboxone®
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Subject's Self Assessment Using 10 cm Visual Analogue Scale (VAS) of Overall Preference for One of the Two Buprenorphine-based Maintenance Therapies (Suboxone® or Subutex®).
Description: Score of 0 = "Not satisfied at all"; Score of 10 = "Totally satisfied"
Time Frame: Each treatment Day (post-dose on days 1-5)
Population: Intent to Treat (ITT) - each day's results were based on number of subjects who had a Day 1 visit.
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Day 1 (Subutex®); Day 2 (Subutex®); Day 3 (Suboxone®); Day 4 (Suboxone®); Day 5 (Suboxone®): All subjects in this trial received Subutex® for first two days of study followed by Suboxone® for last 3 days of study
Arm/Group | Day 1 (Subutex®) | Day 2 (Subutex®) | Day 3 (Suboxone®) | Day 4 (Suboxone®) | Day 5 (Suboxone®)
Number analyzed (Participants) | 53 | 53 | 53 | 53 | 53
centimeters | 7.04 (2.24) | 6.83 (2.18) | 7.38 (1.93) | 6.89 (2.48) | 7.12 (2.26)
Statistical Analysis 1: Comparison: Day 1 (Subutex®) vs Day 2 (Subutex®) vs Day 3 (Suboxone®) vs Day 4 (Suboxone®) vs Day 5 (Suboxone®); Test type: Superiority or Other; p = 0.130, ANCOVA — p-value adjusted for treatment only; Mean Difference (Net) = 0.42 — Difference between treatments (Suboxone minus Subutex)estimated by ANCOVA = 0.42

ADVERSE EVENTS:
Arm/Group | Subutex®/Suboxone®
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 8/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subutex®/Suboxone® (N=53)
Fatigue (General disorders) | 4 (4)
Headache (Nervous system disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor agreement is always necessary before PI publishing or communications. The sponsor can review the communication project during 28 days. The sponsor can require changes to the communication and can extend the embargo.